CLINICAL TRIAL: NCT06614712
Title: A Multinational, Observational, Retrospective, Secondary Data Study Describing Management and Treatment in Routine Clinical Practice Among Patients With Chronic Kidney Disease. Local Adaptation for Spain. Part 1
Brief Title: OPTIMISE-CKD Study_current Clinical Landscape in Spain
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169AR00032
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1: Pre-pricing & reimbursement, incident renal disease cohort (study observation period 2020- 2024)
  Interventions: Other: Pre-pricing & reimbursement, incident renal disease cohort (study observation period 2020- 2024)
- Cohort 2: Post-pricing & reimbursement, incident renal disease cohort (study observation period 2023-2024)
  Interventions: Other: Post-pricing & reimbursement, incident renal disease cohort (study observation period 2023-2024)

INTERVENTIONS:
Other: Pre-pricing & reimbursement, incident renal disease cohort (study observation period 2020- 2024) — Incident renal disease patients in this cohort are defined as those that newly met the renal function measurement definition stated above, with first-ever registered laboratory UACR and/or eGFR measurements or CKD diagnosis on or after the start date of this cohort study period, the 1st August 2020 and until the 1 st February 2023 (DAPA_CKD P&R date in Spain). The first of the dates fulfilling any of the criteria defined above for the renal function measurement or CKD diagnosis, is defined as the patient index date-1 of this study cohort.
  At the index date-1, the renal disease will be staged based on eGFR (and/or UACR measurements in addition, if available) as specified in the KDIGO guidelines.
  Patients will be followed up from the index date-1 until the end of continuous enrolment, last date of available data or date of death, until the end of the overall observation period.
  Groups: Cohort 1
Other: Post-pricing & reimbursement, incident renal disease cohort (study observation period 2023-2024) — We define the post-P&R cohort including all incident renal disease patients observed in the dapagliflozin-CKD post-pricing and reimbursement period. Patients in this cohort newly met the renal function measurement definition stated above, with first-ever registered laboratory UACR and/or eGFR measurements or CKD diagnosis on or after the 1 st February 2023 (DAPA_CKD P&R date in Spain) and until the end of the study observation period. The first of the dates fulfilling any of the criteria defined above for the renal function measurement or CKD diagnosis, is defined as the patient index date-2 of this study cohort. At the index date-2, the renal disease will be staged based on eGFR (and/or UACR measurements in addition, if available) as specified in the KDIGO guidelines. Patients will be followed up from the index date-2 until the end of continuous enrolment, last date of available data or date of death, until the end of the overall study period
  Groups: Cohort 2

SUMMARY:
OPTIMISE-CKD is a retrospective, observational study, using secondary data. The incidence of renal disease, including CKD, using eGFR or UACR laboratory measurements and diagnostic codes will be assessed in the study population. The study will also assess the incidence of selected cardiovascular and renal events and the current use of kidney-protective treatments

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years as of study index date

* With renal function measured as either of the following:

  * At least 1 UACR measure of ≥30 mg/g; OR
  * At least 2 eGFR measures taken ≥90 days apart, of which both eGFR is ≤75 ml/min/1.73m2 ; OR
* registered with Chronic Kidney Disease (CKD) diagnosis in the medical history (without biochemical confirmation)

Exclusion Criteria:

* History of stage 5 CKD, dialysis, organ transplant, type 1 diabetes, or gestational diabetes on or before the start date of the observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The overall study population will consist of adult patients, aged ≥18 years as of study index date, with their renal function measured
Sampling Method: Non-Probability Sample
Enrollment: 91628 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Baseline demographics and clinical characteristics of the two cohorts of the study, pre-P&R and post-P&R cohorts, at their respective index dates. | from the 1st August 2020 to 30th September 2024
Baseline laboratory measures (number of measures per year and their values) of the two cohorts of the study, pre-P&R and post-P&R cohorts, at their respective index dates. | from the 1st August 2020 to 30th September 2024
Concomitant medications, by drug class and specific drugs of interest (proportion of patients with prescription of selected drugs) of the two cohorts of the study, pre-P&R and post-P&R cohorts, at their respective index dates. | Concomitant medications, by drug class and specific drugs of interest (proportion of patients with prescription of selected drugs) of the two cohorts of the study, pre-P&R and post-P&R cohorts, at their respective index dates.
Initiation of kidney-protective treatment (RAASi or SGLT2i or both) among treatment naïve patients in the pre-P&R cohort and post- P&R | from the 1st August 2020 to 30th September 2024
Discontinuation of newly initiated RAASi or SGLT-2i treatment in the two cohorts of the study, pre-P&R and post-P&R cohorts | from the 1st August 2020 to 30th September 2024
Discontinuation of ongoing RAASi and/or SGLT-2i treatment among treated patients (proportion of patients, time to discontinuation) in the two cohorts of the study, pre-P&R and post-P&R cohorts. | from the 1st August 2020 to 30th September 2024

SECONDARY OUTCOMES:
To describe the current clinical landscape among incident renal disease/incident CKD patients and in new initiators of kidney protective treatment- patients during the follow-up period | from the 1st August 2020 to 30th September 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/